CLINICAL TRIAL: NCT01446666
Title: A Prospective Intra-individual Cohort Study to Compare Gadoxetic Acid (Primovist®)-Enhanced Magnetic Resonance Image and Ultrasonography for the Surveillance of Early Stage Hepatocellular Carcinoma in Patients at High-risk
Brief Title: Gadoxetic Acid-MRI Versus Ultrasonography for the Surveillance of Hepatocellular Carcinoma in High-risk Patients
Acronym: PRIUS
Status: Completed | Type: Observational
Sponsor: Asan Medical Center (Other)
Collaborators: Bayer (Industry)
Responsible Party: Principal Investigator, Young-Suk Lim, Professor, Asan Medical Center
Other Study IDs: AMC2011-0587
Record Dates: First submitted 2011-09-17; First posted 2011-10-05 (Estimated); Results first posted 2019-01-14 (Actual); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Cirrhosis of Liver
Keywords: hepatocellular carcinoma; surveillance; gadoxetic acid; MRI
MeSH Terms: conditions — Fibrosis; Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Buffy coat and serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- HCC high-risk group: Patients with liver cirrhosis with the 1-year risk of HCC of 5% or higher
  ; High Risk Index (>=2.33)
  Risk Index = 1.65 (if the prothrombin activity is <=75%) + 1.41 (if the age is 50 years or older) + 0.92 (if the platelet count is <=100x10(3)/mm3) + 0.74 (if the presence of anti-hepatitis C virus [HCV] or hepatitis B surface antigen [HBsAg] is positive).

SUMMARY:
Current practice guidelines recommend surveillance for hepatocellular carcinoma (HCC) in liver cirrhosis patients with ultrasonography (USG) every 6 months. However, with the advancement of cirrhosis, the sensitivity of USG decreases, while the risk for HCC increases. Gadoxetic acid (Primovist®)-enhanced magnetic resonance imaging (MRI) has been demonstrated to be of clinical value for diagnosis of HCC with the detection sensitivity of 90-95%, which is significantly higher than USG. The hypothesis to be proved by this study is as follows; Primovist-MRI should show significantly higher sensitivity compared to USG for the detection of early stage HCC when both of these imaging modalities are used with the interval of 6 months in patients with cirrhosis at high risk of developing HCC.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is currently the third leading cause of cancer-related deaths worldwide. Cirrhosis, particularly when related to viral hepatitis, is the most notable risk factor for HCC and is found in nearly 80-90% of cases.

The stage of disease at the time of diagnosis largely determines the effectiveness of treatment. The treatment of advanced HCC continues to be primarily palliative, with curative options only available for early HCC. Unfortunately, less than 30% of patients are diagnosed early enough to meet criteria for resection, transplantation, or local ablation.

Surveillance strives to detect HCC at an early stage when it is amenable to curative therapy to reduce mortality. Current practice guidelines recommend surveillance of cirrhotic patients with ultrasonography (USG) every 6 months. However, USG has been reported to have a sensitivity of between 65% and 80% when used as a screening test. However, with the advancement of cirrhosis, the sensitivity of USG decreases, while the risk for HCC increases.

Gadoxetic acid (Primovist®)-enhanced magnetic resonance imaging (MRI) of the liver has been demonstrated to be of clinical value for local staging before HCC surgery and for the assessment of patients with inconclusive conventional imaging findings. The detection sensitivity of Primovist-MRI has been known to be as high as 90-95%, which is significantly higher than USG or multiphase computer tomography (CT) scan. MRI does not have radiation exposure, which is a meaningful merit to be used as a surveillance test. However, MRI has never been considered for surveillance or screening of HCC.

Thus, the hypothesis to be proved by this study is as follows; Primovist-MRI should show significantly higher sensitivity compared to USG for the detection of early stage HCC when both of these imaging modalities are used with the interval of 6 months in patients with cirrhosis at high risk of developing HCC. The investigators will also analyze whether the specificity of Primovist-MRI are not compromised by its high sensitivity.

ELIGIBILITY:
Inclusion Criteria:

Patients with liver cirrhosis with the 1 year risk of HCC of 5% or higher meeting all of following criteria;

1. The evidence of cirrhosis of any etiology within 12 months prior to screening Definition of cirrhosis by any of following methods

   * 1) Histologically by liver biopsy;
   * 2) Non-histologically by evidence of portal hypertension in the presence of chronic liver disease;

     * Evidence of portal hypertension, including any of followings;

       1. The identification of splenomegaly on USG, CT, or MRI examinations with typical features of cirrhosis
       2. The identification of esophageal or gastric varices on endoscopic examination
2. High Risk Index (>=2.33); Risk Index = 1.65 (if the prothrombin activity is <=75%) + 1.41 (if the age is 50 years or older) + 0.92 (if the platelet count is <=100x10(3)/mm3) + 0.74 (if the presence of anti-hepatitis C virus [HCV] or hepatitis B surface antigen [HBsAg] is positive).
3. Older than 20 years of age
4. Absence of previous or current history of HCC
5. Absence of HCC should be identified by liver USG, dynamic CT, or contrast-enhanced MRI within 6 months prior to screening
6. Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0-2
7. Patient is able to comply with scheduled visits, evaluation plans, and other study procedures.
8. Patient is willing to provide written informed consent

Exclusion Criteria:

Presence of any of following criteria;

1. Active or suspected cancer other than HCC, or a history of malignancy where the risk of recurrence is >20% within 2 years
2. Child-Pugh score >9
3. Significant medical comorbidities in which survival is predicted to be less than 3 years
4. Estimated glomerular filtration rate (GFR) < 30 mL/min/1.73m2
5. Precautions for MRI (cardiac pacemaker, ferromagnetic implants, etc.)
6. Severe claustrophobia that may interfere with protocol compliance.
7. Any other condition which, in the opinion of the Investigator, would make the patient unsuitable for enrollment or could interfere with the completing the study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospital out-patient clinic
Sampling Method: Non-Probability Sample
Enrollment: 423 (Actual)
Dates: Start 2011-11; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Young-Suk Lim, MD, PhD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Kim HL, An J, Park JA, Park SH, Lim YS, Lee EK. Magnetic Resonance Imaging Is Cost-Effective for Hepatocellular Carcinoma Surveillance in High-Risk Patients With Cirrhosis. Hepatology. 2019 Apr;69(4):1599-1613. doi: 10.1002/hep.30330. Epub 2019 Feb 25. PMID 30365164
- [Derived] Kim SY, An J, Lim YS, Han S, Lee JY, Byun JH, Won HJ, Lee SJ, Lee HC, Lee YS. MRI With Liver-Specific Contrast for Surveillance of Patients With Cirrhosis at High Risk of Hepatocellular Carcinoma. JAMA Oncol. 2017 Apr 1;3(4):456-463. doi: 10.1001/jamaoncol.2016.3147. PMID 27657493

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were recruited between November 2011 and August 2012. The inclusion criteria for participation were an age of 20 years or older and the presence of cirrhosis with an estimated annual HCC risk of >5%.
Pre-assignment Details: The absence of hepatocellular carcinoma (HCC) had been evaluated by US, dynamic CT scan, or MRI within 6 months before enrollment. Patients with Child-Pugh class C liver function or estimated glomerular filtration rate <30 mL/min/1.73m^2 were excluded.
Groups:
- US+MRI: The patients were evaluated by three rounds of screening tests with paired US and gadoxetic acid-enhanced MRI at 6-month intervals
Period: Overall Study
Arm/Group | US+MRI
Started | 407 (Among the 423 participants who consented, 15 withdrew the consent and one died.)
Completed | 326
Not Completed | 81

BASELINE CHARACTERISTICS:
Arm/Group | US+MRI
Number analyzed (Participants) | 407
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 56 [52 to 62]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 177
  Male | 230
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Korean | 407
Region of Enrollment [Count of Participants; unit: Participants]
  South Korea | 407

OUTCOME MEASURES:

1. Primary Outcome: Detection Rate of Patients With HCC
Description: - The number of patients with definite HCC detected by a given modality divided by the total number of patients with definite HCC detected by any of 2 modalities plus interval cancers
Time Frame: during the 1.5-year study period (from the date of first screening to 6 months following the last screening)
Measure: Number; unit: percentage of HCC detected on each exam
Groups:
- Ultasonography: Results from ultrasonography
- Gadoxetic Acid-enhanced MRI: Results from Gadoxetic acid-enhanced MRI
Arm/Group | Ultasonography | Gadoxetic Acid-enhanced MRI
Number analyzed (Participants) | 43 | 43
percentage of HCC detected on each exam | 27.9 | 86.0
Statistical Analysis 1: Comparison: Ultasonography vs Gadoxetic Acid-enhanced MRI; The HCC detection rate was defined as the number of patients with HCC detected by a given modality divided by the total number of patients with HCC detected by all modalities and by follow-up dynamic CT scan. The HCC detection rates from ultrasonography and MRI were compared; Test type: Superiority; p < 0.01, McNemar

2. Secondary Outcome: Detection Rate of Patients With Early Stage HCC
Description: * The number of patients with early stage HCC detected by a given modality divided by the total number of patients with early stage HCC detected by any of 2 modalities plus interval cancers.
  * Early stage (stage A or 0) HCC is defined by the Barcelona Clinic Liver Cancer staging system (BCLC): A single HCC <5 cm or <=3 lesions each <3 cm in diameter, without gross vascular invasion or extrahepatic metastasis.
Time Frame: during the 1.5-year study period (from the date of first screening to 6 months following the last screening)
Measure: Number; unit: percentage of early HCC detected
Arm/Group | Ultasonography | Gadoxetic Acid-enhanced MRI
Number analyzed (Participants) | 42 | 42
percentage of early HCC detected | 26.2 | 85.7
Statistical Analysis 1: Comparison: Ultasonography vs Gadoxetic Acid-enhanced MRI; Test type: Superiority; p < 0.01, McNemar

3. Secondary Outcome: Detection Rate of Patients With Very Early Stage HCC
Description: * The number of patients with HCC nodules of very early stage detected by a given modality divided by the total number of definite HCC nodules of very early stage detected by any of 2 modalities plus interval cancers.
  * Very early stage (stage 0) HCC is defined by the Barcelona Clinic Liver Cancer staging system (BCLC): A single HCC <2 cm without gross vascular invasion or extrahepatic metastasis.
Time Frame: during the 1.5-year study period (from the date of first screening to 6 months following the last screening)
Population: Of the 43 patients, 32 (74.4%) had very early-stage.
Measure: Number; unit: percentage of detected very early HCC
Arm/Group | Ultasonography | Gadoxetic Acid-enhanced MRI
Number analyzed (Participants) | 32 | 32
percentage of detected very early HCC | 27.3 | 84.8
Statistical Analysis 1: Comparison: Ultasonography vs Gadoxetic Acid-enhanced MRI; Test type: Superiority; p < 0.01, McNemar

4. Secondary Outcome: False Positive Rate
Description: The false-positive rate was defined as the number of tests with positive findings by a specific imaging modality in patients without a HCC.
Time Frame: during the 1.5-year study period (from the date of first screening to 6 months following the last screening)
Measure: Number; unit: percentage of false positive test
Units Other Than Participants: the number of exams
Arm/Group | Ultasonography | Gadoxetic Acid-enhanced MRI
Number analyzed (Participants) | 364 | 364
Number analyzed (the number of exams) | 1057 | 1057
percentage of false positive test | 5.6 | 3.0
Statistical Analysis 1: Comparison: Ultasonography vs Gadoxetic Acid-enhanced MRI; Test type: Superiority; p = 0.004, McNemar

5. Secondary Outcome: Positive Predictive Value for HCC
Description: The positive predictive value was the number of true positive test results in patients with the positive tests in a specific modality.
Time Frame: during the 1.5-year study period (from the date of first screening to 6 months following the last screening)
Measure: Number; unit: percentage of true positive calls
Arm/Group | Ultasonography | Gadoxetic Acid-enhanced MRI
Number analyzed (Participants) | 71 | 69
percentage of true positive calls | 16.9 | 53.6

ADVERSE EVENTS:
Arm/Group | US+MRI
Serious Adverse Events (participants affected / at risk) | 0/407
Other Adverse Events (participants affected / at risk) | 0/407

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No